CLINICAL TRIAL: NCT04815005
Title: HoFH, the International Clinical Collaborators - A Global HoFH Data-sharing Platform
Brief Title: HoFH, the International Clinical Collaborators Registry
Acronym: HICC
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Amsterdam (Other); University of Cape Town (Other); University of Witwatersrand, South Africa (Other)
Responsible Party: Sponsor
Other Study IDs: HICC
Record Dates: First submitted 2021-03-04; First posted 2021-03-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Homozygous Familial Hypercholesterolemia
Keywords: Homozygous Familial Hypercholesterolemia; Autosomal Dominant; Hypercholesterolemia; Autosomal Recessive Hypercholesterolemia; Registry
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia; Multiple Pterygium Syndrome, Autosomal Dominant; Hypercholesterolemia; Hyperlipoproteinemia Type III | interventions — Demography; Genotype

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HoFH: Patients diagnosed with HoFH by their physicians, either based on clinical or genetic criteria.
  Interventions: Other: Demographics, diagnosis type, genotype, lipid profile, treatment allocation, country of residence.

INTERVENTIONS:
Other: Demographics, diagnosis type, genotype, lipid profile, treatment allocation, country of residence. — Differences in diagnosis, genotype, lipid profile treatment allocation among HoFH patients worldwide.

SUMMARY:
Homozygous familial hypercholesterolemia (HoFH), a rare inherited disorder caused by bi-allelic mutations in the LDL Receptor pathway, is characterized by extremely elevated levels of low-density lipoprotein cholesterol (LDL-C) from birth and premature atherosclerotic cardiovascular disease (ASCVD). Our current knowledge about HoFH is disjointed and largely stems from relatively small case series and expert opinion. HICC (Homozygous FH International Clinical Collaborators) is a global consortium of clinicians who are contributing de-identified data of patients diagnosed with HoFH with the goal to advance our understanding of this rare disease.

DETAILED DESCRIPTION:
The HICC registry is an observational, multicenter, international registry collecting de-identified clinical and genetic information from patients with homozygous Familial Hypercholesterolemia (HoFH) worldwide.

Patients are eligible to be enrolled in the registry based on the diagnosis of HoFH by the treating clinician, irrespective of how the diagnosis was made. To generate up-to-date data reflecting current rather than historic practice, patients who died or were lost to follow-up prior to 2010 are excluded.

Anonymized data on demographics, type of HoFH diagnosis (clinical and/or based on the results of a genetic test), genetic results, (cardiovascular) medical history, relevant family history, physical examination, laboratory measurements, lipid lowering treatment and cardiovascular imaging are collected for 3 different time points: at diagnosis, at enrolment and at time of best lipid profile (if this is different from time at enrolment). Data are collected using pre-definite electronic case report forms to ensure uniformity of data collected. Primary analysis will be cross-sectional (e.g. based on country of residence, age, etc)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of homozygous familial hypercholesterolemia (HoFH) clinically of genetically determined

Exclusion Criteria:

* No diagnosis of HoFH

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The registry aims to include data from as many patients diagnosed with HoFH as possible. All patients must be living at time of entry into the database or have been deceased within the last 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants entered into the database | Through study completion, an average of 8 years
  Number of study participants with homozygous familial hypercholesterolemia

SECONDARY OUTCOMES:
Untreated and treated LDL-C levels across world income regions | Through study completion, an average of 8 years
  Number of treated versus number of untreated subjects with relevant LDL-C levels

CONTACTS AND LOCATIONS:
Overall Officials: Marina Cuchel, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (4):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States
- Department of Vascular Medicine, Amsterdam UMC, Amsterdam, Netherlands
- South Africa (2):
  - Department of Medicine, Division of Lipidology and Hatter Institute for Cardiovascular Research in Africa, University of Cape Town, Cape Town
  - c. Carbohydrate and Lipid Metabolism Research Unit, Faculty of Health Sciences, University of Witwatersrand, Johannesburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mulder JWCM, Schonck WAM, Tromp TR, Reijman MD, Reeskamp LF, Hovingh GK, Blom DJ, Roeters van Lennep JE. Real-world family planning and pregnancy practices in women with homozygous familial hypercholesterolemia. Atherosclerosis. 2025 May;404:119187. doi: 10.1016/j.atherosclerosis.2025.119187. Epub 2025 Apr 3. PMID 40250039
- [Derived] Tromp TR, Hartgers ML, Hovingh GK, Vallejo-Vaz AJ, Ray KK, Soran H, Freiberger T, Bertolini S, Harada-Shiba M, Blom DJ, Raal FJ, Cuchel M; Homozygous Familial Hypercholesterolaemia International Clinical Collaborators. Worldwide experience of homozygous familial hypercholesterolaemia: retrospective cohort study. Lancet. 2022 Feb 19;399(10326):719-728. doi: 10.1016/S0140-6736(21)02001-8. Epub 2022 Jan 28. PMID 35101175